CLINICAL TRIAL: NCT06713174
Title: Assessment of Interleukin 8 and 10 Level Changes Before and During Root Canal Treatment for Necrotic Pulp with Apical Periodontitis
Brief Title: Interleukin 8 And10 Levels Changes in Teeth with Necrotic Pulp and Apical Periodontitis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Faculty of Dental Medicine for Girls (Other Government)
Responsible Party: Principal Investigator, Esraa Mohamed elsagheer Hassan, Dentist at ministry of health, Faculty of Dental Medicine for Girls
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ENDOD-101-1-b
Record Dates: First submitted 2024-11-25; First posted 2024-12-03 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Pulp and Periapical Tissue Disease; Patients with Pulp Necrosis and Apical Periodontitis
Keywords: interleukin 8; interleukin 10; necrotic pulp; periodontitis
MeSH Terms: conditions — Periapical Periodontitis; Dental Pulp Necrosis; Periodontitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- assessment of interleukin 8,10 pre and post (Other): Gingival crevicular fluid sampling Gingival crevicular fluid (GCF) will be collected at two different time points. The collection periods will be defined as follows: before initiating access into the root canal (period 1), and before canal filling (period 2).
  Periapical Fluid sample:
  Periapical fluid samples will be collected at two different time points. The collection periods will be defined as follows: just after crown access and before root canal filling , by introducing 3 sequential sterile absorbent paper points of a size compatible with the root canal. These paper points will be introduced into the canal until they extend 2 mm beyond the radiographically determined apex.
  Interventions: Diagnostic Test: Assessment of Interleukin 8 and 10 Level Changes Before and During Root Canal Treatment for Necrotic Pulp with Apical Periodontitis

INTERVENTIONS:
Diagnostic Test: Assessment of Interleukin 8 and 10 Level Changes Before and During Root Canal Treatment for Necrotic Pulp with Apical Periodontitis — This study will be performed to investigate interleukin-8 (IL-8) and interleukin-10 (IL-10) level changes in gingival crevicular fluid (GCF) and periapical fluid before and during root canal treatment (RCT) in patients with necrotic pulp and apical periodontitis. The null hypothesis tested will be There is no significant difference in (IL-8) and (IL-10) levels in gingival crevicular fluid (GCF) and periapical before and during root canal treatment (RCT) for necrotic pulp with apical periodontitis.

SUMMARY:
The goal of this observational study is to evaluate changes in interleukin 8 (IL-8) and interleukin 10 (IL-10) levels in gingival crevicular fluid (GCF) and periapical fluid during root canal treatment in patients with necrotic pulp and apical periodontitis. The main question it aims to answer is:

How do IL-8 and IL-10 levels in GCF and periapical fluid change over the course of treatment?

Participants will:

Provide samples of GCF and periapical fluid at two different time points during their root canal treatment.

Undergo treatment based on standard clinical protocols for necrotic pulp and apical periodontitis.

DETAILED DESCRIPTION:
This observational study aims to investigate changes in biomarkers within gingival crevicular fluid (GCF) and periapical fluid during root canal treatment for patients with necrotic pulp and apical periodontitis. Ethical approval was obtained from the Research Ethics Committee (REC) of the Faculty of Dentistry for Girls at Al-Azhar University (P-EN-23-04). Written informed consent will be obtained from all participants after explaining the study's aims and importance.

Study Design:

Patients requiring root canal treatment at the Endodontic Clinic, Faculty of Dental Medicine for Girls, Al-Azhar University, will be recruited based on inclusion and exclusion criteria.

Inclusion Criteria:

Adults aged 18-45 years. Patients without systemic diseases. Patients diagnosed with necrotic pulp and apical periodontitis in a single-rooted tooth with a single canal.

Patients with no previous endodontic treatment or related therapeutic procedures.

Patients with normal periodontal health.

Exclusion Criteria:

Patients who decline participation. Patients on long-term anti-inflammatory medication, immunosuppressive chemotherapy, or antibiotics within the last 3 weeks.

Patients with systemic health conditions (e.g., cardiovascular diseases, diabetes mellitus, HIV, hepatitis).

Pregnant women, smokers, and those with unrestorable teeth.

Sample Collection Procedures:

1. Gingival Crevicular Fluid (GCF):

   Timing: Samples will be collected at two time points:

   Before initiating access into the root canal (Period 1). Before canal filling (Period 2).

   Procedure:

   Isolation of the area using cotton rolls. Plaque removal and gentle air drying of the tooth. Placement of sterilized paper strips in the gingival sulcus until minimal resistance is felt.

   Strips will remain for one minute and will be placed on mesial or distal vestibular surfaces.

   If blood contamination occurs, collection will be attempted from another site. Persistent bleeding will lead to sample exclusion.

   Storage:

   Strips will be placed in Eppendorf tubes with phosphate-buffered saline and frozen at -80°C until analysis.
2. Periapical Fluid:

Timing: Samples will be collected:

Just after crown access. Before root canal filling.

Procedure:

Three sequential sterile absorbent paper points will be inserted into the root canal, extending 2 mm beyond the radiographic apex.

Points will be left undisturbed for one minute. The tips (4 mm) will be cut and placed in Eppendorf tubes containing 2 mL of reduced transport fluid (RTF).

Storage:

Tubes will be stored at -80°C until analysis.

Root Canal Treatment Protocol:

Anesthesia and Isolation:

Local anesthesia with 2% lidocaine containing epinephrine 1:80,000. Rubber dam isolation.

Access and Cleaning:

Access cavity preparation using round tungsten carbide burs. Gates Glidden burs for straight-line access. Cleaning and shaping with stainless steel K-files. Irrigation with 10 mL of 2.5% sodium hypochlorite (total duration: 30 minutes). Final rinse with 2 mL of 17% EDTA for 1 minute, followed by 2 mL of sterile saline.

Sample Collection:

After initial preparation, samples from periapical fluid will be collected as described.

Temporary filling material will be used to seal the access cavity.

Completion of Treatment:

Seven days later, temporary fillings will be removed, and second samples of GCF and periapical fluid will be collected.

The root canals will be filled using gutta-percha and epoxy resin sealer via lateral compaction.

Composite resin will seal the access cavity.

Storage and Analysis:

All samples will be preserved at -80°C until biomarker analysis is performed. The study focuses on evaluating changes in key biomarkers (e.g., interleukins) associated with inflammation and healing during treatment.

This description ensures clarity, technical detail, and adherence to ethical and procedural standards, avoiding duplication of information from other sections

ELIGIBILITY:
Inclusion Criteria:Inclusion Criteria:

1. Adult patients aged between 18 and 45 years.
2. Patients without any systemic diseases.
3. Patients diagnosed with pulp necrosis and apical periodontitis of a single root with a single canal who are seeking endodontic treatment.
4. Patients who have not previously received endodontic treatment or any related therapeutic procedures.
5. Patients with normal periodontal health.

Inclusion Criteria:

1. Adult patients aged between 18 and 45 years. 2. Patients without any systemic diseases. 3. Patients diagnosed with pulp necrosis and apical periodontitis of a single root with a single canal who are seeking endodontic treatment. 4. Patients who have not previously received endodontic treatment or any related therapeutic procedures. 5. Patients with normal periodontal health.

-

Exclusion Criteria:

* Exclusion Criteria:

  1. Patients who refuse to participate in the study.
  2. Patients who have been on long-term anti-inflammatory medication,received immunosuppressive chemotherapy or taken antibiotics within the last 3 weeks.
  3. Patients with systemic health conditions such as cardiovascular and respiratory diseases, diabetes mellitus, HIV infection, or hepatitis.
  4. Unrestorable teeth, pregnant women, and smokers will also be excluded from the study

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Estimated)
Dates: Start 2024-12-15 (Estimated); Primary Completion 2025-01-15 (Estimated); Study Completion 2025-01-30 (Estimated)

PRIMARY OUTCOMES:
To assess changes in IL-8 and IL-10 levels in GCF and periapical fluid and evaluate if they are equivalent and can be used as markers of the inflammatory response before and during RCT. | The study will collect data at various time points, including baseline (pre-RCT) and during RCT.

IPD SHARING:
Plan to Share IPD: No